CLINICAL TRIAL: NCT05068180
Title: Low-dose Neuroleptanalgesia Reduce the Occurrences of Postoperative Delirium in Elderly Patients Undergoing Non-cardiac Major Surgery : a Randomized Controlled Trial
Brief Title: Low-dose Neuroleptanalgesia for Postoperative Delirium in Elderly Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai 8th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY2020-125
Record Dates: First submitted 2021-09-06; First posted 2021-10-05 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Sigmoid Neoplasms; Liver Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Osteoarthropathy; Fractures, Bone; Gynecologic Cancer
Keywords: Postoperative delirium; Neuroleptanalgesia; Aged; Noncardiac major surgery
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Sigmoid Neoplasms; Liver Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Fractures, Bone; Emergence Delirium | interventions — Neuroleptanalgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neuroleptanalgesia group (Experimental): Droperidol 1.25 mg and fentanyl 0.025 mg (diluted with normal saline up to 5ml) is to be administrated intravenously 30 minutes before the end of the procedure.
  Interventions: Drug: low-dose neuroleptanalgesia
- Control group (Placebo Comparator): The same volume of normal saline is to be administrated intravenously 30 minutes before the end of the procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: low-dose neuroleptanalgesia — Droperidol 1.25 mg and fentanyl 0.025 mg (diluted with normal saline up to 5ml) is to be administrated intravenously 30 minutes before the end of the procedure.
  Arms: Neuroleptanalgesia group
Drug: Placebo — The same volume of normal saline is to be administrated intravenously 30 minutes before the end of the procedure.
  Arms: Control group

SUMMARY:
Postoperative delirium（POD）is a common complication that can directly affect important clinical outcomes, and exert an enormous burden on patients, their families, hospitals, and public resources. In order to evaluate whether an intraoperative administration of low-dose neuroleptanalgesia reduces postoperative delirium, droperidol 1.25 mg and fentanyl 0.025 mg or normal saline is used by intravenous injection 30 minutes before the end of the operation, in elderly patients with non-cardiac major surgery under general anesthesia. The efficiency and safety of neuroleptanalgesia on the incidence of POD would be evaluated in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years old and ≤ 85 years old;
2. Selective non-cardiac major surgery;
3. Informed consent and voluntary participation in the trial;
4. ASA class I-II;
5. Anticipated operation duration ≥ 2 hours;
6. No plan to ICU after operation.

Exclusion Criteria:

1. Neurosurgery;
2. Patients with neurological and mental diseases: such as basal ganglia disease, Parkinson's syndrome, severe central nervous depression, Alzheimer's disease , etc;
3. Patients with prolonged Q-T interval, cardiac repolarization disorder and other severe arrhythmia;
4. Patients with severe cardiopulmonary disease, liver and kidney dysfunction;
5. Allergic or contraindications to droperidol or fentanyl citrate;
6. Admitted to ICU after operation.
7. Operation duration < 2 hours;

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-04-10 (Estimated); Study Completion 2022-04-10 (Estimated)

PRIMARY OUTCOMES:
Incidences of POD after general anesthesia in elderly patients undergoing non-cardiac major surgery | Up to 7 days after surgery（or leaving hospital）

SECONDARY OUTCOMES:
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Incidence of postoperative nausea and vomiting | Up to 7 days after surgery（or leaving hospital）
Patients' satisfaction | Up to 7 days after surgery（or leaving hospital）
  This outcome will be measured using a numeric rating scale from 1 ( dissatisfaction ) to 3 (very satisfied)
Incidence of postoperative hypoxia | Up to 1 day after surgery
Incidence of major serious complications and serious arrhythmia | Up to 7 days after surgery（or leaving hospital）
Duration of postoperative delirium | Up to 7 days after surgery（or leaving hospital）

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Doctor, Study Chair — RenJi Hospital
Locations (2):
- China (2):
  - Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Eighth People's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No